CLINICAL TRIAL: NCT07239596
Title: An Open, Multicenter Phase Ib/II Clinical Study of SHR-8068 in Combination With Adebrelimab and Other Anti-tumor Drugs for the Treatment of Advanced Renal Cell Carcinoma
Brief Title: Phase Ib/II Clinical Study of SHR-8068 Combined With Adebrelimab and Other Anti-tumor Drugs in the Treatment of Advanced Renal Cell Carcinom
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Suzhou Suncadia Biopharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHR-8068-207-RCC
Record Dates: First submitted 2025-11-16; First posted 2025-11-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2025-11

CONDITIONS: Advanced Renal Cell Carcinoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- SHR-8068+ Adebrelimab + Bevacizumab (Experimental)
  Interventions: Drug: SHR-8068；Adebrelimab ；Bevacizumab
- SHR-8068+ Adebrelimab +HS-10516 (Experimental)
  Interventions: Drug: SHR-8068；Adebrelimab ；HS-10516
- SHR-8068+ Adebrelimab + Bevacizumab +HRS-10516 (Experimental)
  Interventions: Drug: SHR-8068； Adebrelimab ； Bevacizumab ；HRS-10516

INTERVENTIONS:
Drug: SHR-8068；Adebrelimab ；Bevacizumab — SHR-8068+ Adebrelimab + Bevacizumab
  Arms: SHR-8068+ Adebrelimab + Bevacizumab
Drug: SHR-8068；Adebrelimab ；HS-10516 — SHR-8068+ Adebrelimab +HS-10516
  Arms: SHR-8068+ Adebrelimab +HS-10516
Drug: SHR-8068； Adebrelimab ； Bevacizumab ；HRS-10516 — SHR-8068+ Adebrelimab + Bevacizumab +HRS-10516
  Arms: SHR-8068+ Adebrelimab + Bevacizumab +HRS-10516

SUMMARY:
This study evaluated the safety and efficacy of SHR-8068 in combination with Adebrelimab and other anti-tumor drugs in the treatment of advanced renal cell carcinoma

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 75 years old (including boundary values)
2. Volunteer to participate in this clinical study and sign informed consent;
3. ECOG score 0-1;
4. Expected survival ≥3 months;
5. Patients with locally advanced unresectable or metastatic clear cell renal cell carcinoma confirmed by histology or cytology;
6. Tumor tissue samples must be provided for testing
7. There is at least one measurable or evaluable lesion that meets the RECIST 1.1 criteria;
8. Adequate bone marrow and organ function.

Exclusion Criteria:

1. Have previously used or are currently using HIF inhibitors.
2. Had received chemotherapy, immunotherapy, targeted therapy, anti-tumor traditional Chinese medicine or other clinical research drugs within 4 weeks prior to the first administration of the study; Palliative radiotherapy was received within 2 weeks before the first administration.
3. Live attenuated vaccines are used within a certain period of time before the first medication as stipulated in the plan, or it is expected that such vaccines will be needed during the treatment period.
4. Undergoing major surgical treatment within a certain period of time after the first administration of medication (excluding diagnosis) or expecting major surgical treatment during the study period.
5. There are severe gastrointestinal function abnormalities in clinical practice, which may affect the intake, transportation or absorption of drugs.
6. Suffering from other active malignant tumors within 3 years or at the same time.
7. Patients who have received organ transplants in the past (excluding corneal transplants).
8. A clinically significant thrombotic or embolic event occurred within 6 months prior to the first administration of the drug.
9. There are clinical symptoms or diseases of the heart that are not well controlled.
10. Active tuberculosis.
11. Moderate and severe ascites with clinical symptoms; Uncontrolled or moderate to excessive pleural effusion and pericardial effusion.
12. The toxicity and/or complications of previous intervention measures have not been restored to the level of NCI-CTCAE≤1 or the inclusion and exclusion criteria.
13. Subjects with active hepatitis B or active hepatitis C.
14. As determined by the researcher, there are other factors that may affect the research results or lead to the forced termination of this study midway

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Estimated)
Dates: Start 2026-01-06 (Actual); Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) | 21days after the first administration of each subject
  DLT defined as the Incidence and severity of adverse events
Overall response rate(ORR) | from first dose to disease progression or death, whichever comes first, up to 3 years
  Defined as percentage of participants who achieved a best overall response of complete response (CR) or partial response (PR) assessed by the investigator

SECONDARY OUTCOMES:
Progression-free survival (PFS) by investigator | Until progression or death, assessed up to approximately 3 year
  Defined as time from first administration until progression or death as assessed by the investigator
Duration of response (DOR) by investigator assessment | Until progression or death, assessed up to approximately 3 year
  Defined as the time from the first documented objective response (CR or PR) to the first documented disease progression or death assessed by the investigator
Disease control rate (DCR) by investigator assessment | Until progression, assessed up to approximately 3 year
  Defined as percentage of participants who achieved a best overall response of complete response (CR), partial response (PR) or stable disease (SD) assessed by the investigator
Incidence and severity of adverse events (AEs)/serious adverse events (SAEs) | until to 90 days after the last dose，assessed up to approximately 3 years
  Incidence and severity of adverse events (AEs)/serious adverse events (SAEs) graded by Common Terminology Criteria for Adverse Events (CTCAE) v5.0

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided